CLINICAL TRIAL: NCT01354743
Title: Upper Facial Remodeling With Perlane-L and Dysport.
Acronym: DPL-2010
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beer, Kenneth R., M.D., PA (Individual)
Collaborators: Medicis Pharmaceutical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DysportPerlaneL-2010
Record Dates: First submitted 2011-05-11; First posted 2011-05-17 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-09

CONDITIONS: Mild to Moderate Temporal Atrophy; Moderate to Severe Glabellar Rhytids; Moderate to Severe Periorbital Rhytids
Keywords: atrophy; rhytids; glabellar; periorbital
MeSH Terms: conditions — Atrophy | interventions — abobotulinumtoxinA

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dysport (Other): Dysport injections into the glabella and orbicularis oculi muscles with dose based on muscle mass
  Interventions: Drug: Dysport; Device: Perlane L

INTERVENTIONS:
Drug: Dysport — Patients entering will be based on gender and assessment of procerus and corrugator muscle mass. Muscle mass will be graded separately for males and females as +, ++, or+++ (light/small, moderate/medium, or heavy/large) by assessment of the procerus/corrugator muscles. Male patients will receive 0.3 mL to 0.4 mL (60, 70, or 80 units) in five equally divided doses of Dysport™ Female patients will receive 0.25 mL to 0.35 mL (50, 60 or 70 units) in equally divided doses of Dysport™ at 5 designated injection sites in the glabellar region
  Subjects will be treated with Dysport™ 20 or 30 units bilaterally to crow's feet.
  Subjects will be treated at baseline and if maximum amount of product has not been used at 1 month follow up subject will receive a touch up. No further treatment will be done for the remaining study visits.
Device: Perlane L — The subject will be allowed to receive up to 4 mls between the temporal fossa and the glabella area.

SUMMARY:
The purpose of this study is to provide data to support combination treatment of the upper face with Perlane-L® and Dysport™. This study will assess the outcome of upper face rejuvenation in the temporal fossa; outcome of glabella and/or periorbital regions will also be assessed as a secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient,male or female subjects of any race, 40-75 years of age.
* Mild to Moderate temoral atrophy of (1 or 2 on Four Point Temporal Atrophy Scale)
* One of the following:

Periocular rhytids characterized by a measurement of 3 or more during maximum attempted muscle contraction (during maximum smiling) upon evaluation using the Rao-Goldman 5 point Facial Wrinkle Scale.

Mild to moderate glabella rhytiuds by a measurment of 3 or more upon evaluation using the Rao-Goldman 5-point Facial Wrinkle Scale.

* Subjects will be enrolled if previous history of facial cold sores, but will be medicated to avoid any recurrence.
* able to understand the requirements of the study and sign a Institutional Review Board Informed Consent/HIPPA Authorization forms and receive a copy.
* Subjects of childbearing potential must have a negative urine pregnancy test result at baseline and practice a reliable method of contraception throughout the study: A female is considered of childbearing potential unless she is post menopausal for >12 months prior to study drug administration.
* without a uterus and/or both ovaries; or
* surgically sterile (e.g., tubal ligation) for >6 months prior to study drug administration.

The following methods of contraception, if properly used, are generally considered reliable for females of childbearing potential who may participate in the study:

* hormonal contraceptives† (oral, patch, injection, implant);
* male condom with intra-vaginal spermicide or diaphragm or cervical cap with spermicide;
* vaginal contraceptive ring;
* intrauterine device;
* surgical sterilization (bilateral tubal ligation);
* partner vasectomized††; or
* total sexual abstinence*.

  * Hormonal contraceptives must be started at least 90 days prior to study drug administration, and intra-uterine contraceptive device must be placed at least 30 days prior to study drug administration.

    * Vasectomized >3 months or with a 0 sperm count; * Female subjects of childbearing potential who are not sexually active are not required to practice a reliable method of contraception. They may be enrolled at the Investigator's discretion provided that they are counseled to remain sexually inactive for the duration of the study and understand the possible risks involved in getting pregnant during the study.

Exclusion Criteria:

* Previous injection of botulinum toxin of any serotype within 6 months, Previous injection of semi-permanent fillers in the upper face (i.e. glabella, periorbital, temporal areas) within the last 12 months. Previous injection of permanent fillers in the upper face (i.e. glabella, periorbital, temporal areas) are excluded.
* Subjects who are pregnant (positive urine pregnancy test), breast-feeding, or who are of childbearing potential and not practicing a reliable method of birth control.
* Subjects planning a facial cosmetic procedure during the study period or with prior cosmetic procedures (i.e., surgery) or visible scars that may affect the evaluation of response.
* Facial asymmetry, ptosis, excessive dermatochalasis, deep dermal scarring,thick sebaceous skin, or an inability to substantially lessen upper facial rhytids even by physically spreading them apart.
* Previous cosmetic surgery to the upper face (e.g., periorbital surgery, brow lift, eyelid or eyebrow surgery, etc.).
* Laser resurfacing, or soft tissue augmentation in the periocular area in the 12 months preceding Visit 1.
* Medical condition that may increase their risk of exposure to botulinum toxin including diagnosed Myasthenia Gravis, Eaton-Lambert Syndrome, Amyotrophic Lateral Sclerosis, or any other disease that might interfere with neuromuscular function.
* Current use of aminoglycoside antibiotics, curare-like agents, or agents that might interfere with neuromuscular (skeletal) function.
* Profound atrophy/excessive weakness of muscles in target areas of injection.
* History of facial nerve palsy.
* Any patients with known autoimmune disease or compromised immune systems ie HIV, AIDS or current chemotherapy.
* Infection at the injection site or systemic infection (in this case, postpone study entry until one week following recovery).
* Allergy or sensitivity to any component of Dysport™ and/or Perlane-L®.
* Evidence of recent alcohol or drug abuse.
* Medical and/or psychiatric problems that is severe enough to interfere with the study results (Investigator opinion).
* History of poor cooperation, non-compliance with medical treatment, or unreliability.
* Exposure to an investigational drug study within 30 days of the Baseline Visit.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-12; Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Upper face rejuvenation in the temporal fossa | 9months
  Subjects are assessed from a Four Point Temporal Atropy scale at baseline(must present with a 1 or 2 score).Subject will be assessed at 1 month with additonal treatment if needed and return at month 3,6, and 9 months and be assessed with the Four Point Atrophy Scale.

SECONDARY OUTCOMES:
Measure of rejuvenation in glabella and/or periorbital regions | 9 months
  Mild to moderate glabella rhytids and Periocular rhytids by a measurement of 3 or more upon evaluation using the Rao-Goldman 5-point Facial Wrinkle Scale.
  Subject will be assessed at 1 month with additonal treatment if needed and return at month 3,6, and 9 months and be assessed with Rao-Goldman 5-point Facial Wrinkle Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Beer M.D., Principal Investigator — Kenneth Beer, M.D., PA
Locations (1):
- Kenneth R. Beer, M.D., PA, West Palm Beach, Florida, United States